CLINICAL TRIAL: NCT05347862
Title: Remote and Intensive Program for Physical Activity Promotion for People With Type 2 Diabetes: a Pragmatic Clinical Trial - The PRACTICE Trial
Brief Title: Remote and Intensive Program for Physical Activity Promotion for People With Type 2 Diabetes (The PRACTICE Trial)
Acronym: PRACTICE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Federal University of Rio Grande do Sul (Other); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20210394
Record Dates: First submitted 2022-04-14; First posted 2022-04-26 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-12

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 diabetes mellitus; randomized controlled trial; physical activity; aging; pragmatic clinical trial
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Motor Activity | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: This is a pragmatic trial to assess the effectiveness of a physical activity promotion program on reduction levels of glycated hemoglobin in patients with Type 2 diabetes.
Who Masked: Outcomes Assessor
Masking Description: Single-blind masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Other): Usual standard advice to practice physical activity as an important measure to promote health benefits.
  Interventions: Other: Control group
- Physical Activity Promotion (Experimental): The intervention will consist of telephone calls and text messages to promote the practice of 150 minutes/week of physical activity in the daily life of participants.
  Interventions: Other: Physical activity promotion

INTERVENTIONS:
Other: Control group — At baseline, this group will receive only the usual standard advice to practice physical activity as an important measure to promote health benefits. During the intervention period, they will receive only telephone calls monthly to assess the physical activity practice, changes in medication, and adverse events. When appropriate, evaluations of 12 and 24 weeks will be scheduled.
  Arms: Control group
Other: Physical activity promotion — The intervention will be based on a remote approach, for 24 weeks. The intervention will consist of telephone calls and sent messages to promote the practice of 150 minutes/week of physical activity in the daily life of participants, plus short text messages promoting health behaviors related to self-care, nutrition, physical activity, and sedentary behavior.
  Initially, this group will be followed weekly during the first 4 weeks. After this period this group can up to two weekly calls, according to their preference. The text messages will be weekly. During the telephone calls, the research team will verify the volume of PA achieved and help the participants to identify and overcome barriers to PA practice, and motivate and register any adverse events related or not to the study.
  Arms: Physical Activity Promotion

SUMMARY:
The purpose of this trial is to evaluate the effects of a remote and intensive physical activity promotion program for people with Type 2 Diabetes (T2D), in comparison to a usual model of PA counseling, in glycemic levels, level of physical activity and quality of life in adults in elderly with T2D.

DETAILED DESCRIPTION:
The PRACTICE Trial aims to assess the effectiveness of a remote and intensive physical activity promotion program in contrast to the usual advice for physical activity on the management of HbA1c in people with T2DM.

The duration of the trial will be 24 weeks. Participants will be allocated to the intervention group or control group. The data collection will include variables related to (a) physical activity levels; (b) quality of life; (c) self-care in T2D; (d) functional capacity levels; and (e) adverse events related or not to the study.

ELIGIBILITY:
Inclusion Criteria:

* Eighteen years of age or older;
* Glycated hemoglobin ≥ 8.0%;
* Being a resident in Porto Alegre or metropolitan areas (Viamão, Alvorada, Cachoeirinha, or Canoas);
* Eligibility to perform physical activity after cardiovascular risk assessment;
* Have some means of access to the internet (direct access or via a family member who can receive the research material and share the information/material sent with the participant).

Exclusion Criteria:

* Physically active, that is, performing at least 150 minutes of moderate to vigorous PA per week;
* Not having their own cell phone capable of receiving calls and text messages;
* Progressive neurological disorder (e.g., Parkinsonism, Alzheimer's Disease);
* Psychiatric disorder that makes the intervention unfeasible;
* Physical, language, hearing, vision or cognition disorder that makes it impossible to attend the evaluations and carry out the intervention;
* Severe cardiovascular disease (class III and IV heart failure, unstable angina), history of macrovascular event in the last 12 months (acute myocardial infarction, revascularization procedures, deep vein thrombosis, stroke or pulmonary embolism);
* Joint, muscle or bone injury that makes the intervention unfeasible;
* Planning to move to cities outside the geographic area where the study is carried out;
* Inadequate control of comorbidities. Resting systolic blood pressure >180 mmHg and/or resting diastolic blood pressure >100 mmHg;
* Physical limitation that makes it impossible or brings risk to the participant's practice (e.g. lower limb amputation that makes locomotion difficult, use of crutches, cane).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 344 (Estimated)
Dates: Start 2022-12-02 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Glycated Hemoglobin at 3 and 6 months | Baseline; 12 weeks; 24 weeks.
  Glycated hemoglobin (HbA1c) is the primary outcome used for the comparison of a remote and intensive physical activity promotion program compared with usual advice for physical activity. The minimum clinically important difference considered for the study design and sample size calculation was an HbA1c reduction of 0.50% in favor of the remote and intensive physical activity promotion program.

SECONDARY OUTCOMES:
Physical Activity Levels | Baseline; 12 weeks; 24 weeks.
  The levels of physical activity will be assessed using the International Physical Activity Questionnaire (IPAQ, Portuguese version).
Sitting time | Baseline; 12 weeks; 24 weeks.
  The sitting time will be assessed using the International Physical Activity Questionnaire (IPAQ, Portuguese version).
Medication changes | Monthly, up to 24 weeks.
  Participants' reports of medication changes (increases, decreases, or no changes in medication treatment) during the intervention period.
Short Form Health Survey (SF-36) | Baseline; 12 weeks; 24 weeks.
  This instrument is a self-administered 36-item questionnaire. The score of quality of life ranges from 0 to 100, in which higher scores are indicative of better quality of life.

OTHER OUTCOMES:
Blood pressure | Baseline; 12 weeks; 24 weeks.
  This outcome will be assessed by measuring systolic and diastolic blood pressure in accordance to clinical guidelines and using an automated oscillometric device.
Walking capacity | Baseline; 12 weeks; 24 weeks.
  Total distance (in meters) performed during the six-minute walk test.
Handgrip strength | Baseline; 12 weeks; 24 weeks.
  Maximum strength (in kgf) achieved by both hands in a handgrip test using a hand dynamometer.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Umpierre, PhD, Principal Investigator — Hospital de Clínicas de Porto Alegre
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data after will be shared after trial completion. Data usage will be under the PI's auspices, but restrictions or screenings will not be imposed upon data requests. Outcomes data and any deemed relevant support information (sociodemographic, clinical history and allocated groups) will be shared if available.
  Details regarding the study's design and statistical plan can be obtained consulting the trial's protocol (links to be added as soon as available).
  Data on other outcomes could be requested contacting the PI. Data access will be available after all participants completed the study and will remain accessible for as long as deemed necessary by the study's committee. Data sets, variables' dictionary and statistical analysis description will be made available online upon registration and acceptance of the study team's data sharing terms and policy.
Supporting Information: Study Protocol
Time Frame: The individual participant dataset will become available in a public repository up to six months after the first study publication.
Access Criteria: A simple registration will grant access to study datasets. The website for these files is not defined at the time of registration.

REFERENCES:
- See also: Study repository - Open Science Framework — https://osf.io/npxdw/